CLINICAL TRIAL: NCT00085020
Title: A Phase I, Open-Label Study of the Safety, Tolerability and Pharmacokinetics of GW572016 in Combination With Trastuzumab [Herceptin†]
Brief Title: GW572016 and Trastuzumab in Treating Patients With Metastatic Breast Cancer That Overexpresses HER2/Neu
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000367118; UCLA-0305039; GSK-EGF10023
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; male breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: trastuzumab
Drug: lapatinib ditosylate

SUMMARY:
RATIONALE: GW572016 may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Monoclonal antibodies, such as trastuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Giving GW572016 with trastuzumab may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of GW572016 when given together with trastuzumab in treating patients with metastatic breast cancer that overexpresses HER2/neu.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the optimally tolerated regimen of GW572016 when administered with trastuzumab (Herceptin^®) in patients with metastatic breast cancer that overexpresses HER2/neu.
* Determine the safety and tolerability of this regimen in these patients.

Secondary

* Determine the pharmacokinetic parameters of this regimen in these patients.
* Determine the clinical response in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter, dose-escalation study of GW572016.

Patients receive oral GW572016 once daily on days 1-28 and trastuzumab (Herceptin^®) IV over 90 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of GW572016 until the optimally tolerated regimen (OTR) is determined. The OTR is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the OTR is determined, 10-18 additional patients are entered and treated at the OTR.

Patients are followed at 28 days.

PROJECTED ACCRUAL: A total of 3-35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer
* Metastatic disease
* Measurable or evaluable disease
* HER2/neu overexpression (2+ or 3+) confirmed by immunohistochemistry and/or HER2 gene amplification by fluorescence in situ hybridization
* Brain metastases treated by surgery and/or radiotherapy allowed provided the following criteria are met:

  * Neurologic status stable 2 weeks after discontinuing dexamethasone
  * No concurrent anticonvulsants that induce metabolism (e.g., phenytoin, carbamazepine, or phenobarbital)
* 18 and over
* Male or female
* Karnofsky 70-100%
* Life expectancy, At least 12 weeks
* Hematopoietic

  * Absolute granulocyte count ≥ 1,500/mm^3
  * Platelet count ≥ 100,000/mm^3
  * Hemoglobin ≥ 9 g/dL
  * AST and ALT ≤ 3 times upper limit of normal (ULN) (5 times ULN if patient has liver metastases)
  * Bilirubin < 1.5 mg/dL
  * Creatinine clearance > 30 mL/min
* Cardiovascular

  * LVEF > 50%
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* Adequate venous access
* Able to swallow and retain oral medication
* Prior adjuvant/neoadjuvant chemotherapy allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin.
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior major surgery
* Recovered from all prior therapy
* More than 28 days since prior participation in another investigational study
* More than 28 days since prior investigational drugs

Exclusion Criteria:

* extensive tumor, pleural effusions, or parenchymal masses) resulting in dyspnea at rest
* uncontrolled brain metastases or leptomeningeal disease
* prior myocardial infarction
* pre-existing cardiac dysfunction (e.g., congestive heart failure)
* clinically significant cardiac disease
* angina pectoris
* symptomatic intrinsic pulmonary disease (e.g., asthma or chronic obstructive pulmonary disease) resulting in dyspnea at rest
* pregnant or nursing
* active infection
* known hypersensitivity to Chinese Hamster Ovary cell proteins or any component of this product
* known immediate or delayed hypersensitivity reaction or idiosyncrasy to products of similar chemical composition as study drug
* known contraindications to trastuzumab (Herceptin^®)
* malabsorption syndrome
* disease significantly affecting gastrointestinal function
* psychiatric disorder that would preclude study compliance
* other serious illness or condition
* concurrent biologic therapy
* prior cumulative dose of doxorubicin > 400 mg/m^2 (including liposomal doxorubicin)
* concurrent hormonal therapy*
* concurrent glucocorticoids
* concurrent radiotherapy
* prior major resection of the stomach or small bowel that could affect absorption of GW572016
* concurrent cytotoxic therapy
* other concurrent anticancer therapy
* other concurrent investigational drugs during and for 28 days after study treatment
* concurrent administration of any of the following medications or substances:
* Antibiotics

  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Ciprofloxacin
  * Rifampin
  * Norfloxacin
  * Rifabutin
* HIV antivirals

  * Delaviridine
  * Indinavir
  * Nelfinavir
  * Ritonavir
  * Saquinavir
  * Efavirenz
  * Nevirapine
  * Amprenavir
  * Lopinavir
* Anticonvulsants

  * Phenytoin
  * Carbamazepine
  * Phenobarbital
* Antidepressants

  * Fluoxetine
  * Nefazodone
  * Fluvoxamine
* Antifungals

  * Itraconazole
  * Ketoconazole
  * Fluconazole
  * Voriconazole
* Antacids (within 1 hour before and after study drug administration)
* Cimetidine
* Amiodarone
* Diltiazem
* Pioglitazone
* Hypericum perforatum (St. John's wort)
* Grapefruit or grapefruit juice
* Rifabutin
* Diethyldithiocarbamate
* Gestodene
* Mifepristone
* Modafinil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-03; Primary Completion 2004-12 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Pegram, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Storniolo AM, Burris HA III, Overmoyer B, et al.: A phase I, open-label study of the safety, tolerability and pharmacokinetics of lapatinib (GW572016) in combination with trastuzumab. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-1040, 2005.
- [Result] Burris III HA, Storniolo AM, Overmoyer EA, et al.: A phase I, open-label study of the safety, tolerability and pharmacokinetics of lapatinib (GW572016) in combination with trastuzumab. [Abstract] Breast Cancer Res Treat 88 (1): A-3043, 2004.